CLINICAL TRIAL: NCT04579900
Title: Dissecting Host-microbiome Modifiers of Type 2 Diabetes Risk
Acronym: DBBIOTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, André Marette, Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CMI2 CHU
Record Dates: First submitted 2020-10-06; First posted 2020-10-08 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Type 2 Diabetes patients (Experimental): Upper gut biopsies and lower gut samples
  Interventions: Procedure: Endoscopy and duodenal biopsy and sampling
- Non Type 2 Diabetes patients (Active Comparator): Upper gut biopsies and lower gut samples
  Interventions: Procedure: Endoscopy and duodenal biopsy and sampling

INTERVENTIONS:
Procedure: Endoscopy and duodenal biopsy and sampling — All volunteers will have endoscopy and duodenal biopsy and will have to provide stool samples

SUMMARY:
It is now well documented that changes in gut microbiota composition accompany obesity and type 2 diabetes (T2D) and contribute to low-grade inflammation, insulin resistance,and glucose intolerance. It is not yet clear if T2D predisposes the intestine to allow more microbial products or possibly live bacteria to subvert the gut mucosal barrier. However, it is known that hyperglycemia during T2D induces a more permissive gut barrier allowing increased penetration of microbes and their products into the blood. An important next step is to determine which strains of bacteria promote dysbiosis, allowing bacteria or bacterial components to subvert the gut barrier and alter glucose control. It is hypothesized that gut microbes in the colon and other lower gut segments are key modulators of energy balance, glucose homeostasis and insulin sensitivity.

DETAILED DESCRIPTION:
The gut acts as a barrier to bacteria and nutrients and participates in glucose homeostasis via endocrine actors and the gut-brain-peripheral axis. It is unclear how T2D alters microbes in upper and lower intestine of humans. Studies in animals show that T2D promotes translocation of microbes to the blood and tissues to promote metabolic dysfunction. It is crucial to determine whether bacteria or their components subvert the gut barrier in human T2D, and then to identity the relevant bacterial strains in tissues that control blood glucose. The overall objective of our research program is to demonstrate that specific microbes in the gut, circulation, and key metabolic tissues are involved in the progression of T2D. We will define the microbial signatures of T2D in duodenal biopsies and stool samples by comparing T2D and non-T2D subjects.

ELIGIBILITY:
Inclusion Criteria:

* T2DB de novo or non T2DB patients

Exclusion Criteria:

* oral hypoglycemic agents or lipidlowering or antihypertensive drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-02-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Microbial signature | One week
  Compare the bacterial profile of T2D and non-T2D subjects

CONTACTS AND LOCATIONS:
Overall Officials: André Marette, PhD, Principal Investigator — Laval University
Locations (1):
- INAF, Université Laval, Québec, Quebec, Canada